CLINICAL TRIAL: NCT05559593
Title: War Impact on the Final Year Ukrainian Resident's Competence Acquisition
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Assistant professor at the Department of OF SURGERY, ANESTHESIOLOGY AND INTENSIVE THERAPY OF POSTGRADUATE EDUCATION, Bogomolets National Medical University
Other Study IDs: HJ45kds32
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Educational Problems
Keywords: medical education; anaesthesiology; war

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study to identify the war impact on the second (final) year residents-anaesthesiologists' education quality and their ability to get necessary competencies.

DETAILED DESCRIPTION:
The study was conducted at the postgraduate surgery, anesthesiology and intensive care department of Bogomolets National Medical University (Bogomolets NMU).

It started before the war to assess the education quality and residents-anesthesiologists readiness for independent work after two years of residency. When the war started, the study was continued and then results 2021 compared against 2022.

In Ukraine we have a 2-year residency program in anaesthesiology and intensive care, it includes 12 months of a so-called theoretical part, which is provided by postgraduate faculties with rotation on different clinical departments of the faculty (like obstetric anaesthesiology, cardio anaesthesiology, intensive care, transplantology, thoracic anesthesiology etc.), and 10 months of practical part - in one of the major acute hospitals. When Russia invaded Ukraine, 41 final-year residents were studying at the postgraduate department of surgery, anesthesiology and intensive care at Bogomolets NMU. From the 5th day of the war education program was changed to online-based, including an interactive platform for distance learning, ZOOM-meeting for lectures and seminars, and individual work with teachers through online messengers and video calls. 30 (73%) residents and 3 (20%) teachers left Kyiv for 1,5-2 months due to the direct attack of the artillery, missile and troops, with occupied and destroyed Kyiv suburbs, where part of them was living. Those residents, who have left Kyiv, were distributed to hospitals in the Western part of Ukraine to continue their practice in anesthesiology and intensive care departments. Residents, who stayed in Kyiv, were distributed to trauma and military hospitals, which had a lot of patients due to the ongoing war in the city.

After Ukrainian counter offences and Russian withdrawal from the Kyiv district, most of the residents (39) and all teachers came back in April 2022. As a result, live practical sessions and master classes were restored to overtake the program, although we continued online learning with lectures, seminars and other activities.

On the 22nd of June, all residents had an OSCE exam. After passing the OSCE exam, investigators send questionaries' to all residents to reflect on the education quality, competence acquisition and readiness to work as an independent anesthesiologist.

Other questionaries' were sent to all teachers to assess the educational outcomes and war impact, efficacy of the different types of learning and reflection on what needs to be improved.

ELIGIBILITY:
Inclusion Criteria:

* residents-anesthesiologists of the second year

Exclusion Criteria:

* residents-anesthesiologists, who didn't pass final exams

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: residents-anesthesiologists in the second year of postgraduate surgery, anesthesiology and intensive care department of Bogomolets National Medical University
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Educational outcomes evaluation by the final year residents | 2 years
  Educational outcomes evaluation by the final year residents (theoretical and practical parts)

SECONDARY OUTCOMES:
Readiness to work independently in different clinical situations | 2 years
  Readiness of the residents to work independently in different clinical situations.

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, PhD, Study Director — Bogomolets National Medical University
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain N, Panag DS, Srivastava M, Mohan S, Chodnekar SY, Akbari AR, Raj D, Kravarioti D, Swiatek D, Platos E, Khetsuriani K, Gristina KL, Evangelou K, Lica M, Thirumushi RS, Rozani S, Jain S, Fedirko P, Reinis A, Pilmane M. Fate and future of the medical students in Ukraine: A silently bubbling educational crisis. Med Educ. 2022 Aug;56(8):779-782. doi: 10.1111/medu.14818. Epub 2022 May 18. PMID 35502145
- [Background] Raleigh C, Linke A, Hegre H, Karlsen J. Introducing ACLED-armed conflict location and event data. J Peace Res. 2010;47(5):651-660
- [Background] "Ukraine: civilian casualty update 1 August 2022". Office of the United Nations High Commissioner for Human Rights. 1 August 2022. Retrieved 1 August 2022
- [Background] Roland, Gérard. (2006). The Long Run Impact of Bombing Vietnam. Journal of Development Economics. 96. 1-15. 10.1016/j.jdeveco.2010.07.004.
- [Background] Dobiesz VA, Schwid M, Dias RD, Aiwonodagbon B, Tayeb B, Fricke A, Pham P, Erickson TB. Maintaining health professional education during war: A scoping review. Med Educ. 2022 Aug;56(8):793-804. doi: 10.1111/medu.14808. Epub 2022 Apr 25. PMID 35388529
- [Background] UNESKO Institute for Statistics " The quantitative impact of conflict on education". 2011.